CLINICAL TRIAL: NCT04361903
Title: COVID-19: Ruxolitinib for the Treatment of cytokinE Storm resPiratory dIstREss Syndrome. RESPIRE Study
Brief Title: Ruxolitinib for the Treatment of Acute Respiratory Distress Syndrome in Patients With COVID-19 Infection
Acronym: RESPIRE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Azienda USL Toscana Nord Ovest (Other)
Collaborators: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government); Azienda Ospedaliera Universitaria Senese (Other); Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Enrico Capochiani, MD Hematologist, Azienda USL Toscana Nord Ovest
Other Study IDs: 2020.COVID-19.RUXO106
Record Dates: First submitted 2020-04-14; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2
Keywords: Ruxolitinib; Acute Respiratory Distress Syndrome; COVID-19
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19 | interventions — ruxolitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with ruxolutinib: SARS-CoV-2 COVID-19 patients with rapid worsening of respiratory parameters in the last 12 hours treated with ruxolutinib, dosage of at least 20 mg x 2 / day in the first 48 hours.
  Interventions: Drug: Ruxolitinib Oral Tablet

INTERVENTIONS:
Drug: Ruxolitinib Oral Tablet — Ruxolitinib Oral Tablet dosage of at least 20 mg x 2 / day in the first 48 hours

SUMMARY:
It is an observational, cohort, retrospective, monocentric, non-profit study. The primary objective is to evaluate the efficacy and safety of ruxolitinib in acute respiratory distress syndrome in patients with SARS-CoV-2 COVID-19 with rapid deterioration of respiratory parameters in the last 12 hours.

DETAILED DESCRIPTION:
It is an observational, cohort, retrospective, monocentric, non-profit study. Patients with SARS-CoV-2 COVID-19 pneumonia who started off-label Ruxolitinib treatment in the period between 25/03/2020 and 07/04/2020 in hospitalization in the COVID-19 wards of the USL Toscana Nord Ovest company.

Primary objective

- Evaluation of the efficacy and safety of ruxolitinib in acute respiratory distress syndrome in patients with SARS-CoV-2 COVID-19 with rapid deterioration of respiratory parameters in the last 12 hours.

Secondary objectives

* Improvement of respiratory performance.
* Improvement of acute phase inflammation indices.
* Evaluation of known adverse events related to the use of the drug.
* Evaluation of the epidemiological parameters in COVID-19 patients.
* Monitoring of plasma levels of cytokines before and after treatment. Exploratory objectives
* Analysis of the outcomes for the launch of a study on the efficacy and safety of Ruxolitinib in the treatment of ADRS in COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* positive analysis for RT PCR (Shanghai BioTec or Sansure Biotech) for SARS-CoV-2 in a respiratory tract sample;
* Imaging (CT / ECO / RX) positive for pneumonia;
* Oxygen saturation (SaO2) of 93% or less in the environment;
* Partial oxygen pressure ratio (PaO2) on inspired oxygen fraction (FiO2) (PaO2 / FiO2) lower than 250 mg / Hg, but not lower than 100 mg / Hg;
* Rapid clinical evolution with worsening of respiratory parameters in the last 12 hours.
* Release of informed consent.

Exclusion Criteria:

* Pregnancy and breastfeeding;
* Patients already in assisted breathing with tracheal cannula;
* Patients with active and uncompensated serious pathologies previously to the COVID 19 infection;
* Known hypersensitivity to ruxolitinib or to any of the excipients listed in section 6.1 of the SPC;
* Patients with renal insufficiency;
* Patients with positive quantiferon;
* Patients with documented uncontrolled bacterial sepsis (excluding procalcitonin increase in the presence of negative blood cultures);
* Patients with neutropenia equal to or less than 1000 PMN / mmc;
* Patients with thrombocytopenia equal to or less than 100000 / mmc.
* HCV and / or HBV positive patients, HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with SARS-CoV-2 COVID-19 pneumonia who started off-label ruxolitinib treatment in the period between 03/24/2020 and 07/04/2020, with a dosage of at least 20 mg x 2 / day in the first 48 hours
Sampling Method: Non-Probability Sample
Enrollment: 13 (Estimated)
Dates: Start 2020-04-25 (Estimated); Primary Completion 2020-05-24 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients who avoid mechanical assisted ventilation in acute respiratory distress syndrome in patients with SARS-CoV-2 COVID-19 | 15 days
  Number of patients who avoid mechanical assisted ventilation in acute respiratory distress syndrome in patients with SARS-CoV-2 COVID-19 with rapid deterioration of respiratory parameters in the last 12 hours

SECONDARY OUTCOMES:
Improvement of respiratory performance - Arterial Blood Gas Analisys - pH | 15 days
  ABG (arterial Blood Gas): pH as SI Unit, every 12 hours and in any case in the presence of significant clinical variations.
Improvement of respiratory performance - Arterial Blood Gas Analisys - pO2 | 15 days
  ABG (arterial Blood Gas): pO2 in mm Hg, every 12 hours and in any case in the presence of significant clinical variations.
Improvement of respiratory performance - Arterial Blood Gas Analisys - pCO2 | 15 days
  ABG (arterial Blood Gas): pCO2 in mm Hg, every 12 hours and in any case in the presence of significant clinical variations.
Improvement of respiratory performance - ratio values | 15 days
  PaO2 / FiO2, SatO2 ratio. Vital parameters and respiratory function every 12 hours and in any case in the presence of significant clinical variations.
Evaluation of known adverse events related to the use of the drug - D-Dimer | 15 days
  every 24 hours D-Dimer value in mgr/ml
Evaluation of known adverse events related to the use of the drug - fibrinogen | 15 days
  every 24 hours fibrinogen value in mg/dl
Evaluation of known adverse events related to the use of the drug - transaminases | 15 days
  every 24 hours transaminases value in U/L
Evaluation of known adverse events related to the use of the drug - aPTT | 15 days
  every 24 hours aPTT value in seconds
Evaluation of known adverse events related to the use of the drug - INR | 15 days
  every 24 hours INR value in %
Evaluation of known adverse events related to the use of the drug - glycemia | 15 days
  every 24 hours glycemia value in mg/dl
Evaluation of known adverse events related to the use of the drug - creatinine | 15 days
  every 24 hours creatinine serum value in mg/dl
Evaluation of known adverse events related to the use of the drug - Leucocytes count | 15 days
  Total leucocyte as CBC x10e)/L
Evaluation of known adverse events related to the use of the drug - Leucocytes formula | 15 days
  formula % on total leucocyte
Evaluation of the epidemiological parameters: Chest CT | 15 days
  Thoracic imaging, every 48 h: presence, extension and dimension on lung thickening - Chest CT at start and end of treatment, Time elapsed between the onset of clinical symptoms and hospitalization.
Evaluation of the epidemiological parameters: Eco Chest | 15 days
  Thoracic imaging: every day: presence and number of line B every 48 hours.Time elapsed between the onset of clinical symptoms and hospitalization.
Evaluation of the epidemiological parameters: CHEST X-ray | 15 days
  Thoracic imaging: presence, extension and dimension on lung thickening - Chest X-ray, Time elapsed between the onset of clinical symptoms and hospitalization.
Monitoring of Serum levels of cytokines before and every 48 h from start to to end of treatment | 15 days
  Monitoring of serum cytokines (IL-6 in pgr/dL, TNF in pgr/dL) every 48 h
Monitoring incidence of treatment Emergent Adverse Events of ruxolitinib therapy | 15 days
  Number of AE grade 1 to 4

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Dr Capochiani, hematologist, Principal Investigator — Azienda USL Toscana Nord Ovest

REFERENCES:
- [Derived] Capochiani E, Frediani B, Iervasi G, Paolicchi A, Sani S, Roncucci P, Cuccaro A, Franchi F, Simonetti F, Carrara D, Bertaggia I, Nasso D, Riccioni R, Scolletta S, Valente S, Conticini E, Gozzetti A, Bocchia M. Ruxolitinib Rapidly Reduces Acute Respiratory Distress Syndrome in COVID-19 Disease. Analysis of Data Collection From RESPIRE Protocol. Front Med (Lausanne). 2020 Aug 4;7:466. doi: 10.3389/fmed.2020.00466. eCollection 2020. PMID 32850921